CLINICAL TRIAL: NCT02753322
Title: Training Dual-task Balance and Walking in People With Stroke: a Randomized Controlled Trial
Brief Title: Training Dual-task Balance and Walking in People With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Queen Elizabeth Hospital (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, POON Margaret Wai Yee, Senior Physiotherapist, The Queen Elizabeth Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KC/KE-15-0185/ER-3
Record Dates: First submitted 2016-04-24; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Stroke
Keywords: Dual task training; Dual task interference; Sub-acute stroke; Physiotherapy training; Community ambulation; Balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dual-task training group (Experimental): Subjects in this group will have 30 minutes of dual-task training with simultaneously performing balance and walking exercise and attention demanding tasks, and 30 minutes of stretching exercises.
  The training program will last for 8 weeks with frequency of 2 sessions a week.
  Interventions: Other: Dual task training
- Single-task training group (Active Comparator): Subjects in this group will have single-task training with 30 minutes of balance and walking exercise and 30 minutes of attention demanding task performed separately.
  The training program will last for 8 weeks with frequency of 2 sessions a week.
  Interventions: Other: Single-task training
- Limbs exercise group (Active Comparator): Subjects in this group will have stretching and strengthening exercise for 60 minutes.
  The training program will last for 8 weeks with frequency of 2 sessions a week.
  Interventions: Other: Limbs exercise

INTERVENTIONS:
Other: Dual task training — Balance and walking exercises with simultaneously engaging in attention demanding tasks
  Arms: Dual-task training group
Other: Single-task training — Balance and walking exercises and and attention demanding task performed separately
  Arms: Single-task training group
Other: Limbs exercise — Stretching and strengthening exercises
  Arms: Limbs exercise group

SUMMARY:
Stroke is one of the most common chronic disabling conditions in Hong Kong. People after stroke may suffer from certain degree of physical impairment and disability. Resuming safe ambulation in the community appears to be a big challenge to them as it always involves the simultaneous performance of two or more tasks (dual task) such as walking and talking with someone, walking and recalling the shopping list etc. Numerous studies has demonstrated that the interference from dual tasks (dual task interference) may significantly impact the recovery of the functional walking. To date, the relevance of dual task walking to daily community is widely documented and the ability of managing dual task is therefore particularly important. Evidences supported that dual task training showed its promising effect on the balance and walking performance amongst people with neurological disorders, such as chronic stroke. In light of this, the introduction of dual task based balance and walking training into physiotherapy program for stroke patient may enhance the balance and walking performance and hence promote successful community ambulation. Yet, there is limited evidence on its effect in sub-acute stroke.

Objective: To examine the effectiveness of a dual-task based balance and walking training program on performance and dual task interference in balance and walking ability, balance self-efficacy and incidence of falls in people with sub-acute stroke

DETAILED DESCRIPTION:
An assessor-blind, randomized control trial will be conducted. Eighty-four people with sub-acute stroke and fulfill the eligibility criteria will be recruited from the medical wards of the Queen Elizabeth Hospital (QEH) or from the Physiotherapy Department of the QEH. Subjects will be randomly allocated into either dual-task training (DT) group (n=28) or single-task training (ST) group (n=28) or Control (C) group (n=28) by 1:1:1 randomization sequence after baseline evaluation. All subjects will receive usual physiotherapy training. Subjects in the DT group will undergo 30 minutes of dual task training with simultaneously performing balance and walking exercise and attention demanding tasks, and 30 minutes of stretching exercises whereas those in the ST group will undergo single task training with 30 minutes of balance and walking exercise and 30 minutes of attention demanding task performed separately. Subjects in the control group will receive stretching and strengthening exercise only. The training program will last for 8 weeks with frequency of 2 sessions a week and duration of 60 minutes per session.

The degree of the dual-task interference, the balance and walking performance in dual task conditions will be evaluated at three time points: (1) Baseline (within one week before the intervention (2) within one week after completion of training (3) 8 weeks after the completion of training by blinded assessors. Also, the subjects will have monthly telephone follow up on the fall incidence for 6 months after completion of the program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a stroke confirmed by the individual's physician, between 1 month and 6 months post-stroke onset
* Aged ≥50
* Community-dwelling prior to stroke onset (defined as living in one's own home or the home of a relative, friend or caregiver)
* Medically stable
* Montreal Cognitive Assessment (MoCA) scored ≥21
* Ability to follow 3-step commands
* Having motor impairment in the affected lower extremity [Chedoke McMaster Stroke Assessment (CMSA) leg and foot summative score of 4-13 out of 14)], and upper extremity (CMSA arm and hand summative score of 4-13 out of 14)
* Having balance deficits (Mini-Balance Evaluation Systems test score <24)
* Able to ambulate without physical assistance of another person as determined during the 10-meter walk test

Exclusion Criteria:

* Recurrent stroke
* Having neurological conditions other than stroke
* significant receptive and expressive aphasia
* Severe and uncorrected hearing or visual deficits
* Serious musculoskeletal (e.g. amputation) or cardiovascular conditions affecting the ability to exercise (e.g. congestive heart failure), pain experienced at rest or movement, and other serious illnesses that preclude participation.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Degree of the dual-task interference | Baseline, 8 weeks, 16 weeks
  It will be assessed by calculating the percentage of the difference between single task performance (2 walking tasks and 2 balance tasks) and dual task performance of the 2 walking tasks and 2 balance tasks while engaging in 3 attention demanding tasks.

SECONDARY OUTCOMES:
Standing balance with eyes opened in dual task conditions | Baseline, 8 weeks, 16 weeks
  It will be evaluated by Smart Balance System (NeuroCom International Inc., Clackamas, USA). An equilibrium score will be obtained.
Standing balance with eyes closed in dual task conditions | Baseline, 8 weeks, 16 weeks
  It will be evaluated by Smart Balance System (NeuroCom International Inc., Clackamas, USA). An equilibrium score will be obtained.
10 metre walk test in dual task conditions | Baseline, 8 weeks, 16 weeks
  Subjects will be requested to walk along a 14-meter walkway at a self-selected speed. Time taken for the intermediate 10 meters will be recorded.
Obstacle crossing test in dual task conditions | Baseline, 8 weeks, 16 weeks
  Subjects will be asked to walk at their fastest safe speed to cross seven 4-cm-high obstacles along a 10 meters-walkway. Time taken to complete the task will be recorded.
Chinese version of Activities-specific Balance Confidence (ABC) Scale | Baseline, 8 weeks, 16 weeks
  Evaluating the subject's balance self efficacy
Chedoke Arm and Hand Activity Inventory (short form) | Baseline, 8 weeks, 16 weeks
  Performance-based measure for upper limb function
Incidence of falls | From baseline to 6 months
  Fall incidence will be recorded using log book and monthly telephone calls

CONTACTS AND LOCATIONS:
Overall Officials: Margaret WY POON, MSc, Principal Investigator — The Queen Elizabeth Hospital
Locations (1):
- Queen Elizabeth Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No